CLINICAL TRIAL: NCT02228512
Title: Phase I/II Study of Pomalidomide Combined With Modified DA-EPOCH and Rituximab in KSHV-Associated Lymphomas (Primary Effusion Lymphoma and Large Cell Lymphoma Arising in KSHV-Associated Multicentric Castleman Disease)
Brief Title: Study of Pomalidomide Combined With Modified DA-EPOCH and Rituximab in KSHV-Associated Lymphomas
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140176; 14-C-0176
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2015-05-05

CONDITIONS: Large Cell Lymphoma Arising in KSHV-associated Multicentric Castleman Disease; Primary Effusion Lymphoma
Keywords: HHV8; PEL; Immune Modulation; CC-4047; IMiD
MeSH Terms: conditions — Lymphoma, Primary Effusion | interventions — pomalidomide; Rituximab; Prednisone; Etoposide; Doxorubicin; Vincristine; Cyclophosphamide

ARMS (3):
- 1 (Active Comparator): Treatment naive PEL (main cohort)
  Interventions: Drug: Pomalidomide; Drug: Rituximab; Drug: Prednisone; Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide
- 2 (Active Comparator): Treatment na(SqrRoot) ve large cell lymphoma arising in KSHV-MCD
  Interventions: Drug: Pomalidomide; Drug: Rituximab; Drug: Prednisone; Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide
- 3 (Active Comparator): Previously treated KSHV-NHL
  Interventions: Drug: Pomalidomide; Drug: Rituximab; Drug: Prednisone; Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pomalidomide — Part A: 5 mg po daily for 21 days (full course) Part A: 5 mg po daily for 4 days (short course) Part B: 5 mg po daily for 5 days (Phase I/II dose) Part C: Phase I/II dose) po daily Day 1-21 of 28 day cycle for up to 12 cycles.
Drug: Rituximab — Part A: 375 mg/m2 day 22 (full course) Part A: 375 mg/m2 day 5 (short course) Part A: 375 mg/m2 day 1 (omit pomalidomode) Part B: 375 mg/m2 day 1
Drug: Prednisone — Part B: 60 mg/m2/day po x 5 days (day 1-5
Drug: Etoposide — Part B: 50 mg/m2/day CIVI over 24 hrs x 4 days
Drug: Doxorubicin — Part B: 10 mg/m2/day CIVI over 24 hrs x 4 days
Drug: Vincristine — Part B: 0.4 mg/m2/day CIVI over 24 hrs x 4 days
Drug: Cyclophosphamide — Part B: 750 mg/m2 Day 5

SUMMARY:
Background:

- The chemotherapy combination DA-EPOCH-RP includes the drugs etoposide (E), prednisone (P), vincristine (O), cyclophosphamide (C), doxorubicin (H), rituximab (R), and pomalidomide (P). Researchers want to see if including pomalidomide will help people with two rare lymphomas.

Objectives:

- To study the safety and efficacy of the chemotherapy drugs DA-EPOCH-RP.

Eligibility:

- Adults at least 18 years old. They must have primary effusion lymphoma or large cell lymphoma arising from Kaposi sarcoma Herpesvirus-associated multicentric Castleman disease.

Design:

* Participants will be with screened with blood tests, scans, spinal tap, and bone marrow sample. They may have skin or lymph node samples taken and fluid removed from around some organs.
* Participants will have breathing and eye tests. A camera may take pictures inside their body.
* Participants will take pomalidomide alone by mouth for up to 21 days. Then they will get rituximab by intravenous (IV) catheter, which is a small tube that goes into a vein..
* Participants will have an IV inserted in an arm or chest vein to get the IV chemotherapy drugs, at the same time the will take pomalidomide by mouth for 5 days.
* They will get DA-EPOCH-RP in 21-day cycles. Most people will have 6 cycles.
* They will get 4 study drugs by IV for 5 days and 2 others by mouth for 5 days.
* They will get daily filgrastim injections in the skin until white blood counts are acceptable
* For 2 days of some cycles, methotrexate will be injected into the spinal fluid.
* After completing EPOCH-RP, some participants who have Kaposi sarcoma will be prescribed pomalidomide for 3-weeks, followed by a one week break, for up to 12 months.
* Participants will repeat the blood tests often. They will also have repeated medical history, physical exam, urine and stool tests, and pictures of any rashes associated with these lymphomas.
* Participants will have several follow-up visits over 4 years.

DETAILED DESCRIPTION:
Background:

* Kaposi sarcoma herpesvirus (KSHV)-associated primary effusion lymphoma (PEL) and large cell lymphoma arising from KSHV-MCD are aggressive B cell neoplasms with clinicopathologic and molecular profiles distinct from other AIDS-related lymphomas.
* There are no prospective studies on these rare lymphomas. Clinical experience is limited; however, reported prognosis is poor, with median survival estimated at less than 6 months using conventional CHOP-like chemotherapy.
* Novel treatment is urgently needed for KSHV-associated lymphomas, and the therapeutic approach must take into account concurrent KSHV-associated malignancies which are commonly seen in this patient population
* Pomalidomide, an immune-modulatory derivative (IMiD) of thalidomide has in vitro

direct antitumor effect in KSHV-lymphomas as well as immune modulatory and antiangiogenic effects that may be beneficial in treating both KSHV-NHL and in many patients, concurrent KS.

* Rituximab, an anti-CD20 monoclonal antibody, has recently been shown to be an active agent in the management of KSHV-MCD. Although PEL is a CD20-negative tumor, advances in the understanding the biology of KSHV-infection of B-cells, the pathobiology of IL-6 syndromes in KSHV-MCD and KSHV-NHL, and clinical experience using rituximab in the treatment of KSHV-MCD support use of rituximab in the treatment of KSHV-NHL, especially in patients with concurrent KSHV-MCD.
* Modified dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin (DA)-EPOCH is an anthracycline-based regimen that allows for personalization of dose-intensity showing that inclusion of etoposide and infusional administration decreases tumor cell resistance.
* The use of DA-EPOCH in combination with rituximab for the treatment of HIVassociated diffuse large B-cell lymphoma or Burkitt lymphoma has been shown to be safe and effective.
* Given the central role of controlling HIV viremia with combination antiretroviral therapy (cART) in the management of KSHV-associated malignancies, as well as the likely contribution of uncontrolled HIV viremia to PEL pathogenesis, cART will be employed as an important part of the treatment regimen.

Objectives:

Phase I:

-Determine the maximum tolerated dose and/or recommended phase II dose of pomalidomide in combination with DA-EPOCH-R.

Phase II

-Evaluate overall survival in treatment-naive patients with primary effusion lymphoma treated with pomalidomide in combination with, DA-EPOCH and rituximab (DAEPOCH- RP).

Eligibility:

-Adult patients greater than or equal to 18 years with pathology confirmed primary effusion lymphoma,

including extracavitary variant OR large cell lymphoma arising in the setting of KSHVassociated MCD.

* Lymphoma that is measurable or assessable
* Previously treated patients will be allowed if they have not been treated with modified DA-EPOCH or pomalidomide for KSHV-associated lymphoma
* Any HIV status
* Hematologic and biochemical parameters within pre-specified limits at baseline
* Willing to use effective birth control, as defined in the full protocol
* Neither pregnant nor breast feeding
* Excluded if other serious co-morbid condition that would prohibit administration of planned chemotherapeutic intervention is present

Design:

* This is a phase I/ II study of pomalidomide in combination with modified DA-EPOCH-R in patients with PEL and diffuse large cell lymphoma arising in the setting of KSHVMCD.
* Phase I of the study will evaluate escalating doses of pomalidomide (3 mg, 4 mg, and 5 mg) in combination with modified DA-EPOCH-R to determine safe and tolerable phase II pomalidomide dose for combination.
* Treatment in both Phase I and Phase II will have three parts. Patients will receive up to 21 days of pomalidomide monotherapy (part A), followed by 6 cycles of pomalidomide in combination with modified DA-EPOCH-R (part B), and then an optional up to 12 months of pomalidomide (part C) for patients with concurrent KS, symptomatic KSHVMCD, or KSHV inflammatory cytokine syndrome (KICS).
* Patients with HIV will generally be prescribed cART.
* In phase I, with 3 dose levels, 9-18 patients will be accrued (3-6 patients per level).
* In the phase II portion of the study, 15 evaluable patients will be enrolled over 48-60 months and 12 months follow-up after the last patient has enrolled, a 1-tailed 0.10 alpha level test would have 80% power to determine if OS curve would demonstrate a 1-year OS consistent with 45% or better and ruling out 20% or worse.

ELIGIBILITY:
* INCLUSION CRITERIA:

2.1.1.1 KSHV-associated non-Hodgkin lymphoma, with pathology reviewed and confirmed at the NIH. May include WHO recognized tumors

:

2.1.1.1.1 Primary effusion lymphoma (PEL), including extracavitary variant

2.1.1.1.2 Large cell lymphoma arising in the setting of KSHV-associated MCD.

2.1.1.2 Measurable or assessable lymphoma

2.1.1.3 Any HIV status

2.1.1.4 Age 18 years or greater. Because no dosing or adverse event data are currently available on the use of pomalidomide in combination with EPOCH-R in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.

2.1.1.5 ECOG performance status 0-4.

2.1.1.6 Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 14 days prior to and again within 24 hours before starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control

2.1.1.7 All study participants must agree to be registered into the mandatory POMALYST REMS program, and be willing and able to comply with the requirements of the POMALYST REMS program.

2.1.1.8 Able to take aspirin 81mg orally daily or if intolerant of aspirin, able to take a substitute thromboprophylaxis such as low molecular weight heparin.

2.1.1.9 Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

2.1.2.1 Use of other systemic anticancer treatments or agents within the past 2 weeks (4 weeks if the therapy was a monoclonal antibody)

2.1.2.2 Prior dose-adjusted EPOCH or pomalidomide for treatment of KSHV-associated lymphoma

2.1.2.3 Parenchymal brain involvement with lymphoma

2.1.2.4 History of malignant tumors other than KS or KSHV-associated MCD, unless: In complete remission for greater than or equal to 1 year from the time response was first documented or

* Completely resected basal cell carcinoma or
* In situ squamous cell carcinoma of the cervix or anus

2.1.2.5 Inadequate renal function, defined as calculated or estimated creatinine clearance < 60 mL/min unless lymphoma related

2.1.2.6 Inadequate hepatic function:

--2.1.2.6.1 Bilirubin (total) > 1.5 times the upper limit of normal; AST and/or ALT > 3 times the upper limit of normal; EXCEPTIONS:

* Total bilirubin greater than or equal to 5 mg/dL in patients with Gilbert's syndrome as defined by >80% unconjugated
* Total bilirubin greater than or equal to 7.5 with direct fraction > 0.7 if patient is receiving a protease inhibitor at the time of initial evaluation
* Hepatic dysfunction attributed to lymphoma

2.1.2.7 ANC <1000/mm3 and platelets < 75,000/mm3 unless lymphoma, KSHV-MCD, or KICS- related.

2.1.2.8 CTCAEv4.0 Grade 3-4 neuropathy

2.1.2.9 Ejection fraction less than 40% by echocardiography

2.1.2.10 Known drug-related, inherited, or acquired procoagulant disorder including prothrombin gene mutation 20210, antithrombin III deficiency, protein C deficiency, protein S deficiency and antiphospholipid syndrome but not including heterozygosity for the Factor V Leiden mutation or the presence of a lupus anticoagulant in the absence of other criteria for the antiphospholipid syndrome.

2.1.2.11 History of hypersensitivity reactions attributed to thalidomide, lenalidomide, or pomalidomide, including prior development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, lenalidomide, or pomalidomide.

2.1.2.12 Breast feeding (if lactating, must agree not to breast feed while taking pomalidomide). Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Pomalidomide, breastfeeding should be discontinued if the mother is treated with Pomalidomide.

2.1.2.13 Uncontrolled severe intercurrent illness including, but not limited to: bacterial, fungal, or life-threatening viral infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; or psychiatric illness/social situations that would limit compliance with study requirements.

2.1.2.14 Any condition, including laboratory abnormalities, which in the opinion of the Principal Investigator or Lead Associate Investigator, would prohibit administration of planned chemotherapeutic intervention, places the subject at unacceptable risk if they were to participate in the study or confounds the ability to interpret data from the study

2.1.2.15 Pregnant women are excluded from this study because pomalidomide is a Category X agent with the potential for teratogenic or abortifacient effects. These potential risks may also apply to other agents used in this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08-15; Primary Completion 2015-05-05 (Actual); Study Completion 2015-05-05 (Actual)

PRIMARY OUTCOMES:
(Phase I) To determine the maximum tolerated dose and/or recommended phase II dose of pomalidomide in combination with DA-EPOCH-R. | one-year

SECONDARY OUTCOMES:
(Phase II) Evaluate overall survival in treatment naive patients with primary effusion lymphoma treated with pomalidomide in combination with modified DA-EPOCH-RP | one-year
Evaluate response rates and progression free survival | one-year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas S Uldrick, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Dupin N, Diss TL, Kellam P, Tulliez M, Du MQ, Sicard D, Weiss RA, Isaacson PG, Boshoff C. HHV-8 is associated with a plasmablastic variant of Castleman disease that is linked to HHV-8-positive plasmablastic lymphoma. Blood. 2000 Feb 15;95(4):1406-12. PMID 10666218
- [Background] Nador RG, Cesarman E, Chadburn A, Dawson DB, Ansari MQ, Sald J, Knowles DM. Primary effusion lymphoma: a distinct clinicopathologic entity associated with the Kaposi's sarcoma-associated herpes virus. Blood. 1996 Jul 15;88(2):645-56. PMID 8695812
- [Background] Cesarman E, Chang Y, Moore PS, Said JW, Knowles DM. Kaposi's sarcoma-associated herpesvirus-like DNA sequences in AIDS-related body-cavity-based lymphomas. N Engl J Med. 1995 May 4;332(18):1186-91. doi: 10.1056/NEJM199505043321802. PMID 7700311